CLINICAL TRIAL: NCT05479487
Title: Fluzoparib Combined With Apatinib Versus Fluzoparib for Maintenance Treatment in Platinum-Sensitive Relapsed Ovarian Carcinoma: A Randomized, Open Label, Controlled, Multicenter Trial
Brief Title: Fluzoparib and Apatinib Versus Fluzoparib in Relapsed Ovarian Carcinoma Maintenance Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaohua Wu MD (Other)
Responsible Party: Sponsor-Investigator, Xiaohua Wu MD, Professor, Director of Gynecologic Oncology, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-OC-II-005
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Relapsed Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluzoparib+Apatinib combination (Experimental)
  Interventions: Drug: Fluzoparib+Apatinib
- Fluzoparib Monotherapy (Active Comparator)
  Interventions: Drug: Fluzoparib Monotherapy

INTERVENTIONS:
Drug: Fluzoparib+Apatinib — Fluzoparib 100mg bid+ Apatinib 375mg qd
  Arms: Fluzoparib+Apatinib combination
Drug: Fluzoparib Monotherapy — Fluzoparib 150mg bid
  Arms: Fluzoparib Monotherapy

SUMMARY:
This study is a Phase II randomized, open label, controlled, multicenter study to access the effects and tolerability of fluzoparib combined with apatinib versus fluzoparib monotherapy for maintenance treatment in platinum-sensitive relapsed ovarian carcinoma (including patients previous treated with a PARP inhibitor).

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined the study and signed the informed consent
2. Patients ≥18 years of age.
3. Participant has histologically confirmed diagnosis of high-grade predominantly serous ovarian cancer, fallopian tube cancer, primary peritoneal cancer; ≥grade II ovarian endometrioid adenocarcinoma.

   * Mixed mullerian: contain high-grade serous component or endometrioid components over 50%.
4. Participant has received 2 or 3 previous lines of platinum-containing therapy and the last chemotherapy course contains platinum regimen.

   * Preoperative neoadjuvant chemotherapy and postoperative chemotherapy were considered as 1 line chemotherapy treatment.
5. Patient defined as platinum sensitive after this treatment; defined as disease progression greater than 6 months (184 days) after completion of their last dose of platinum chemotherapy
6. Participant has responded to last the platinum regimen (complete or partial response), remains in response and is enrolled on study within 8 weeks of completion of the last platinum regimen.

   * The last chemotherapy must be a platinum-based chemotherapy regimen.
   * Patient must have received at least 4 cycles of treatment for the last platinum-based chemotherapy.
   * A detectable lesion or CA-125 ≥2 ×ULN is required before the last platinum treatment
   * The imaging results showed CR or PR during the last platinum-containing regimen. CA125 decreased to within the ULN or ≥90% from pre-treatment level during treatment and CA125 remained <1xULN or did not increase by >10% in 7 days before the first treatment.
   * If no lesion is assessed prior to chemotherapy, CA125 should be alleviated to the ULN during treatment and maintained at <1xULN for 7 days prior to the first treatment.
7. Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, as assessed within 10 days prior to enrollment.
8. Participant had prior treatment with PARP inhibitor in a maintenance setting:

   * For the BRCA1/2 cohort, the duration of first PARPi exposure must have been ≥18 months following a first line of chemotherapy or ≥12 months following a second line of chemotherapy.
   * For the non BRCA1/2 cohort, the duration of first PARPi exposure must have been ≥12 months following a first line of chemotherapy or ≥6 months following a second line of chemotherapy.
9. Participant has adequate organ function as defined in the following contents (Any blood component or cell growth factor within 14 days prior to randomization is not permitted) Absolute neutrophil count (ANC) ≥1.5×109/L Platelets ≥100×109/L Hemoglobin ≥10g/dL Serum albumin ≥3g/dL Total bilirubin ≤1.5 ×ULN AST (SGOT) and ALT (SGPT) ≤3 × ULN Serum creatinine ≤1.5 × ULN
10. Patients with potential fertility need to use a medically approved contraceptive (such as an intrauterine device, birth control pill or condom) during and for 3 months after the study period; Serum HCG or urine HCG must be negative within 72 hours prior to study enrollment; must be a non-lactation period.

Exclusion Criteria:

1. Prior malignancy unless curatively treated and disease-free for > 5 years prior to study entry. Prior adequately treated non-melanoma skin cancer, in situ cancer of the cervix or breast cancer without recurrence over 3 years allowed.
2. Untreated and/or uncontrolled brain metastases.
3. Not able to swallow pills normally, or have abnormal gastrointestinal function affecting drug absorption as judged by the researcher.
4. Intestinal obstruction within 3 months.
5. The urine protein ≥ ++ and 24-hour urine protein level > 1.0g.
6. Patients with clinical symptoms of cancer ascites, pleural effusion, who need to drainage, or who have undergone ascites drainage within 3 months prior to the first administration;
7. Uncontrolled heart clinical symptoms or diseases, such as :(1) NYHA 2 or more heart failure, (2) Unstable angina pectoris, (3) myocardial infarction within 1 year, (4) Ventricular arrhythmias requiring intervention, (5) QTc>470ms.
8. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds), bleeding tendency or receiving thrombolytic therapy are allowed to receive low-dose low-molecular weight heparin or oral aspirin preventive anticoagulant therapy during the study.
9. Significant bleeding symptoms or clear bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer or vasculitis, etc., within the first 3 months of the randomization. If fecal occultation blood is positive at baseline, gastroscopy should be performed if still positive after reexamination.
10. Active ulcers, unhealed wounds or fractures.
11. Uncontrolled hypertension by antihypertensive medication (systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg).
12. Any bleeding event with grade 2 or higher in CTCAE 5.0 within 4 weeks prior randomization.
13. Active infection or unexplained fever >38.5 degrees during screening or before first treatment.
14. Known to be human immunodeficiency virus positive; Known active hepatitis C virus, or known active hepatitis B virus.
15. Received radiotherapy, chemotherapy, hormone therapy, or molecular targeted therapy, less than 4 weeks after the completion of the last dose or less than 5 drug half-lives before the study for oral molecular targeted drug; Adverse events caused by previous treatment (except hair loss) and not recover to ≤1 degree (CTCAE 5.0).
16. Arteriovenous thrombosis events, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. occurred within 6 months.
17. History of hereditary or acquired bleeding or coagulation disorders (e.g., hemophilia, coagulopathy, thrombocytopenia, etc.).
18. Need receive other systemic anti-tumor therapy during the study period.
19. Other factors that may cause the study to be terminated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) in previous PARP inhibitor treated relapsed ovarian cancer patients. | Up to 2 years
  To determine the efficacy by progression free survival (PFS) of the maintenance treatment in previous PARP inhibitor treated platinum-sensitive relapsed ovarian cancer patients according to RECIST v1.1 criteria (Investigator determined).

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in relapsed ovarian patients | Up to 2 years
  To determine the efficacy by progression free survival (PFS) of the maintenance treatment in platinum-sensitive relapsed ovarian cancer patients according to RECIST v1.1 criteria (Investigator determined).
Progression Free Survival (PFS) in BRCA1/2 mutated relapsed ovarian cancer patients. | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
Disease Control Rate (DCR） | Up to 2 years
Duration of Response (DoR) | Up to 2 years
Overall survival (OS） | Up to 2 years
Adverse Events (AEs) | From the first drug administration to within 30 days for the last treatment dose
  Assese the safety and tolerability of Fluzoparib combined with apatinib maintenance in platinum sensitive relapsed ovarian cancer patients by record the number of participants with of AEs and SAEs, and the proportion of patients with AEs and SAEs, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wu, Ph.D., MD, Principal Investigator — Department of Gynecologic Oncology, Fudan University Shanghai Cancer Center, 270 Dong-An Road, Shanghai 200032, China.

IPD SHARING:
Plan to Share IPD: No
Data is available per require after approved by ethics broad